CLINICAL TRIAL: NCT06226883
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of 3 Active Dose Regimens of MORF-057 in Adults With Moderately to Severely Active Crohn's Disease (GARNET)
Brief Title: A Phase 2 Study to Evaluate MORF-057 in Adults With Moderately to Severely Active Crohn's Disease
Acronym: GARNET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Morphic Therapeutic, Inc. (A Wholly Owned Subsidiary of Eli Lilly and Company) (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 27383; J6E-MC-KWAB (Other: Eli Lilly and Company); MORF-057-203 (Other: Morphic Therapeutic, Inc); U1111-1297-7265 (Other: UTN); 2023-508158-24 (Other: EU Trial (CTIS))
Record Dates: First submitted 2024-01-16; First posted 2024-01-26 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Inflammatory Bowel Diseases; Crohn's Disease
Keywords: Crohn's disease (CD); Inflammatory bowel disease (IBD); a4b7; Moderate-to-severe; Integrin; GARNET
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1 (Part A) (Experimental): Blinded MORF-057 Dosing Regimen 1 for Induction Period and open-label MORF-057 for Maintenance Period
  Interventions: Drug: MORF-057
- Group 2 (Part A) (Experimental): Blinded MORF-057 Dosing Regimen 2 for Induction Period and open-label MORF-057 for Maintenance Period
  Interventions: Drug: MORF-057
- Group 3 (Part A) (Placebo Comparator): Blinded matching placebo for Induction Period and open-label MORF-057 for Maintenance Period
  Interventions: Drug: Placebo; Drug: MORF-057
- Group 4 (Part B) (Experimental): Blinded MORF-057 Dosing Regimen 1 for Induction Period and open-label MORF-057 for Maintenance Period
  Interventions: Drug: MORF-057
- Group 5 (Part B) (Experimental): Blinded MORF-057 Dosing Regimen 2 for Induction Period and open-label MORF-057 for Maintenance Period
  Interventions: Drug: MORF-057
- Group 6 (Part B) (Placebo Comparator): Blinded matching placebo for Induction Period and open-label MORF-057 for Maintenance Period
  Interventions: Drug: Placebo; Drug: MORF-057

INTERVENTIONS:
Drug: Placebo — Matching placebo (identical appearance to MORF-057) administered orally.
  Arms: Group 3 (Part A); Group 6 (Part B)
Drug: MORF-057 — MORF-057 is a small molecule that is designed to selectively inhibit integrin α4β7 and is administered orally.

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled, multicenter study to evaluate the efficacy and safety of 3 active dose regimens of MORF-057 in adult study participants with moderately to severely active Crohn's disease (CD).

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled, multicenter study to evaluate the efficacy and safety of induction therapy with 3 active dose regimens of MORF-057 versus matching placebo in adult study participants with moderately to severely active CD. After completion of the 14-week Induction Period, all participants will receive open-label MORF-057 during the 38-week Maintenance Period. All participants who complete the full 52-week Treatment Period will also have the opportunity to continue treatment in a 52-week Long-Term Extension.

ELIGIBILITY:
Key Inclusion Criteria:

* Has signs/symptoms of CD for at least 90 days prior to screening
* Has a CDAI score of 220 to 450, with an average daily stool subscore ≥4 points and/or an average daily abdominal pain subscore of ≥2 points
* Has an SES-CD score of ≥6 (or an SES-CD score of ≥4 if CD is isolated to the ileum)
* Demonstrated an inadequate response, loss of response, or intolerance to at least one of the following treatments: Corticosteroids, Immunosuppressants (eg, azathioprine, 6-mercaptopurine, methotrexate) and/or advanced therapies for CD (eg, biologic agents, Janus kinase [JAK] inhibitors, applicable investigational products)

Key Exclusion Criteria:

* Diagnosed with indeterminate colitis, microscopic colitis, ischemic colitis, radiation colitis, or UC, or has clinical findings suggestive of UC
* Has CD that is isolated to the oral cavity, stomach, duodenum, jejunum, or perianal region, without colonic or ileal involvement
* Has had extensive bowel resection (>100 cm), and/or more than 3 resections, and/or has a known diagnosis of short bowel syndrome
* Is currently receiving total parenteral nutrition, tube feeding, or a formula diet
* Has positive findings on a subjective neurological screening questionnaire
* Has a concurrent, clinically significant, serious, unstable comorbidity
* Previous treatment with vedolizumab or other licensed or investigational integrin inhibitors
* Is currently participating in any other interventional study or has received any investigational therapy within 30 days
* Previous exposure to MORF-057 and/or a known hypersensitivity to drugs with a similar mechanism to MORF-057
* Unable to attend study visits or comply with study procedures
* Has a history of any major neurological disorders, including: stroke, multiple sclerosis, brain tumor, demyelinating, or neurodegenerative disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with endoscopic response at Week 14 as determined using the Simple Endoscopic Score-CD (SES-CD) | Baseline to Week 14
  The SES-CD is an endoscopic scoring system for evaluating CD activity. Endoscopic response is defined as an SES-CD decrease from baseline of ≥50%

SECONDARY OUTCOMES:
Proportion of participants with clinical response at Week 14 as determined using the Crohn's Disease Activity Index (CDAI) | Baseline to Week 14
  The CDAI is a composite of subscores for clinical and laboratory findings, and patient-reported CD symptoms. Clinical response is defined as a reduction from baseline CDAI score by ≥100 points or a CDAI score of <150 points.
Proportion of participants with clinical remission at Week 14 as determined using the CDAI. | Baseline to Week 14
  The CDAI is a composite of subscores for clinical and laboratory findings, and patient-reported CD symptoms. Clinical remission is defined as a CDAI score of <150 points.

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (160):
- United States (10):
  - Gastro Care Institute, Lancaster, California
  - Wake Research Associates, Raleigh, North Carolina
  - Palmetto Gastroenterology Clinical Research, Summerville, South Carolina
  - Gastrointestinal Associates of Northeast Tennessee, Johnson City, Tennessee
  - GI Alliance - Cedar Park, Cedar Park, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Texas Digestive Disease Consultants, San Marcos, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Care Access Research - Ogden, Ogden, Utah
  - Gastroenterology Associates of Central Virginia, Lynchburg, Virginia
- Austria (4):
  - Medical University Hematology, Innsbruck
  - Salzburg Regional Hospital, Salzburg
  - University Hospital St. Poelten, Sankt Pölten
  - Medical University of Vienna, Vienna
- Brazil (3):
  - Chronos Pesquisa Clínica, Brasília
  - Pesquisare, Santo André
  - Clínica Hepatogastro JK, São Paulo
- Canada (6):
  - Nova Scotia Health Authority, Halifax
  - London Health Sciences Centre, London
  - Diex Recherche Quebec Inc., Québec
  - Mount Sinai Hospital, Toronto
  - St Joseph'S Health Centre Toronto, Toronto
  - Toronto Digestive Disease Associates, Inc., Vaughan
- Colombia (6):
  - Cardiomet Cequin S.A.S., Research Unit, Armenia
  - Fundación Valle del Lili, Cali
  - Cardiovascular Foundation of Colombia, Floridablanca
  - Corporation for Health Studies "CES", Medellín
  - Hospital Pablo Tobon Uribe, Medellín
  - Northern University Foundation Hospital, Soledad
- Croatia (5):
  - Poliklinika Borzan, Osijek
  - Specialty hospital Medico Rijeka, Rijeka
  - Virovitica General Hospital, Virovitica
  - General Hospital Zadar, Zadar
  - Poliklinika Solmed, Zagreb
- Czechia (4):
  - SurGal Clinic s.r.o., Brno
  - Military Hospital Brno,, Brno
  - Clinoxus s.r.o., Outpatient Clinic Budejovicka, Prague
  - Axon Clinical, s.r.o., Prague
- France (3):
  - Hospices Civils de Lyon - Lyon Sud, Pierre-Bénite
  - CHU de Saint-Etienne, Saint-Etienne
  - CHRU Nancy Brabois - Hôpital d'Enfants, Vandœuvre-lès-Nancy
- Georgia (6):
  - High Technology Hospital Medcenter LLC, Batumi
  - Emergency Cardiology Center by Academician G. Chapidze LLC, Tbilisi
  - LTD Institute of Clinical Cardiology, Tbilisi
  - LTD Aversi Clinic, Tbilisi
  - LEPL The First University Clinic of Tbilisi State Medical University, Tbilisi
  - LTD The First Medical Center, Tbilisi
- Germany (9):
  - Charite - University Hospital Berlin, Berlin
  - emovis GmbH - Futuremeds, Berlin
  - DRK Clinic Berlin-Koepenick, Berlin
  - Medical Care Unit Dachau, Dachau
  - Sana Hospital Duisburg, Duisburg
  - University Hospital Halle (Saale), Halle
  - Universitätsklinikum Heidelberg, Heidelberg
  - University Hospital Schleswig-Holstein, Kiel
  - Group Practice Jakobeit, Wipperfürth
- Hungary (6):
  - Bekes Megyei Kozponti Korhaz Dr. Rethy Pal Tagkorhaz IV. Belgyogyaszat, Békéscsaba
  - Semmelweis Medical University, Budapest
  - Markhot Ferenc Oktatókórház, Eger
  - Bugat Pal Hospital Gyongyos, Gyöngyös
  - CLINFAN Szolgáltató Kft, Szekszárd
  - Fejer County St. Gyorgy University Teaching Hospital, Székesfehérvár
- India (13):
  - Navneet Memorial Hospital SUSHRUSHA, Ahmedabad
  - Apollo Cancer Centre, Chennai
  - SMS Medical College Hospital, Jaipur
  - S R Kalla Memorial Gastro and General Hospital, Jaipur
  - Lisie Hospital, Kochi
  - Amrita Institute of Medical Sciences and Research Centre, Kochi
  - Max Super Speciality Hospital, New Delhi
  - Noble Hospital Pvt Ltd, Pune
  - Prime Institute of Digestive Sciences, Rajkot
  - Shree Giriraj Multispeciality Hospital, Rajkot
  - Yashoda Hospital, Secunderabad
  - SIDS Hospital and Research Centre, Surat
  - Samvedna Hospital, Varanasi
- Italy (8):
  - Policlinico S. Orsola-Malpighi, Bologna
  - Big Metropolitan Hospital Niguarda Regional Health Authority, Milan
  - IRCCS San Raffaele, Milan
  - Ospedale Sacro Cuore Don G. Calabria, Negrar
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - IRCCS Istituto Clinico Humanitas- Centro Malattie Infiammatorie Intestinali, Rozzano
  - IRCCS Policlinico San Donato, San Donato Milanese
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Japan (15):
  - Asahikawa Medical College Hospital, Asahikawa
  - Institute of Science Tokyo Hospital, Bunkyō
  - Fukuoka University Chikushi Hospital, Chikushino-shi
  - Kokikai Tsujinaka Hospital Kashiwanoha, Kashiwa-shi
  - Kobe University Hospital, Kobe
  - Yamanashi Prefectural Central Hospital, Kofu
  - Nagasaki University Hospital, Nagasaki
  - Nara Prefecture General Medical Center, Nara
  - Osaka Metropolitan University Hospital, Osaka
  - Saga University Hospital, Saga
  - Tokitokai Tokito Clinic, Saitama
  - Saitama Medical Center, Saitama-Ken
  - Toho University Sakura Medical Center, Sakura
  - Sapporo Higashi Tokushukai Hospital, Sapporo
  - Tokyo Yamate Medical Center, Tokyo
- Kazakhstan (7):
  - Scientific Research Institute of Cardiology and Internal Disease of the Ministry of Health of the Republic of Kazakhstan, Almaty
  - National Research Medical Center, Astana
  - Sana Clinic, Astana
  - Karaganda Medical University, Karaganda
  - Semey Medical University, Semey
  - "Gastromed" Medical Center, Shymkent
  - Diagnostic Center of Shymkent, Shymkent
- Latvia (2):
  - Liepaja Regional Hospital, Liepāja
  - Pauls Stradins Clinical Univeristy Hospital, Riga
- Mexico (8):
  - Applied Neuroscience Research Institute A.C., Durango
  - Proactive CR México SA de CV, Irapuato
  - Medical Clinical Surgical Center Specialized in Research, Jalisco
  - Key Stone Clinical Trials, Mexico City, Distrito Federal
  - Medical Care and Research SA de CV, Mérida
  - Centro de Investigacion Clinica Chapultepec S.A. de C.V., Morelia
  - Oaxaca Site Management Organization, Oaxaca City
  - Centro de Estudios Clínicos de Querétaro (CECLIQ), Querétaro
- Poland (23):
  - "MEDIS" Medical Center, Bydgoszcz
  - Non-public Health Care Center KERmed Medical Centre, Bydgoszcz
  - CLINSANTE Clinical Research Centre Ewa Galczak-Nowak, Malgorzata Trzaska, Bydgoszcz
  - Synexus Polska Sp. Z o.o. Branch in Czestochowa, Częstochowa
  - St. John Paul 2nd Municipal Hospital in Elblag, Elblag
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk
  - Synexus Polska - Katowicach, Katowice
  - "Vita Longa" Non-Public Healthcare Facility, Limited Liability Company, Katowice
  - PLEJADY Medical Centre, Krakow
  - "Landa" Specialist Doctor's Offices, Krakow
  - Twoja Przychodnia Medical Centre of Opole, Opole
  - EMC Medical Institute Joint Stock Company, "Certus" Private Healthcare Facility Hospital No. 1, Poznan
  - Twoja Przychodnia Medical Centre of Poznan, Poznan
  - Synexus Polska Sp. z o.o. Branch in Poznan, Poznan
  - Endoskopia Sp. z.o.o., Sopot
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - H-T. Medical Center, Tychy
  - MDM Healthcare Centre, Warsaw
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - WSD Medi, Warsaw
  - WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Synexus Polska Sp. z o.o., Wroclaw
  - Medical Centre Oporow, Wroclaw
- Romania (4):
  - "Sfanta Vineri" Medical Center, Bucharest
  - Monza Oncology Hospital SRL, Bucharest
  - Colentina Clinical Hospital, Bucharest
  - Oncohelp Association, Timișoara
- Serbia (8):
  - Zvezdara University Medical Center, Belgrade
  - Clinical Center " Dr Dragisa Misovic Dedinje", Belgrade
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - General Hospital Leskovac, Leskovac
  - Clinical Center of Vojvodina, Novi Sad
  - General Hospital Uzice, Užice
  - General Hospital "Djordje Joanovic", Zrenjanin
- Slovakia (4):
  - Cliniq s.r.o., Bratislava
  - ENDOMED s.r.o., Košice
  - GASTRO I., s.r.o., Prešov
  - Gastro LM s.r.o., Prešov
- Spain (6):
  - Complejo Hospitalario Universitario de Ferrol (CHUF)- Hospital Naval, Ferrol
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Universitario Virgen Macarena, Seville
  - University and Polytechnic Hospital La Fe, Valencia